CLINICAL TRIAL: NCT00639080
Title: Necessity for Lipid Lowering Therapy in Type 2 Diabetes Patients
Status: Completed | Type: Observational
Sponsor: Endocrine Research Society (Other)
Responsible Party: Dr. Hugh Tildesley, Endocrine Research Society
Other Study IDs: Necessity for LLT
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2009-08

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Entire study population: All study subjects.
  Interventions: Other: Stop lipid lowering therapy (statin)

INTERVENTIONS:
Other: Stop lipid lowering therapy (statin) — Subjects will only be included in the study and thus asked to stop the statin if they are taking less than or equal to 10 mg of lipitor or an equivalent of another statin.

SUMMARY:
Purpose:

To assess prior need for lipid lowering therapy in patients with type 2 diabetes.

Background/Hypothesis:

At present, lipid lowering therapy, usually with a HMG-CoA reductase inhibitor or "statin", is recommended therapy for selected patients with type 2 diabetes mellitus (DM). The use of statins for primary prevention of CVD is not clear. Some primary prevention studies have found a statistically significant benefit but others have not (CARDS and ASPEN).

Although low-density lipoprotein (LDL) has traditionally been a key marker of cardiovascular disease risk (CVD) risk and thus a guide to statin treatment, in recent years apolipoprotein B (apoB) has emerged as an independent risk factor for CVD.

In a recent study, Tildesley H. et al. showed that in 500 patients with type 2 DM not on lipid lowering therapy there was discordance between LDL and apoB values. Specifically, it was found that among patients who fail to achieve the LDL-C target, 13% of men, 24% of women less than 50 and 13% of women greater than 50 meet the apoB target. In other words, while the LDL level would indicate treatment, the apoB level would not.

Objectives:

The investigators propose to measure lipid parameters during lipid lowering therapy and compare this with lipid parameters at one and two months after discontinuation of therapy in selected patients with type 2 DM at low risk for CVD. Lipid parameters to be measured include: high-density lipoprotein (HDL) - cholesterol, LDL-cholesterol, triglycerides, total cholesterol, total cholesterol: HDL-cholesterol ratio and apoB. As well, A1C will be measured.

ELIGIBILITY:
Inclusion Criteria:

* LDL < 2.5 mmol/L and total cholesterol: HDL-cholesterol ratio < 4.0
* Blood pressure ≤ 130/80 mmHg
* No personal or family history of CVD
* No history of proteinuria or renal failure
* Taking atorvastatin (lipitor) with a dosage ≤ 10 mg, equivalent dosages for other statins follow this requirement (Simvastatin ≤ 20 mg, pravastatin ≤ 40 mg, rosuvastatin ≤ 5 mg, fluvastatin ≤ 40 mg and lovastatin ≤ 40 mg)
* Calculated by the UKPDS Risk Engine to be low risk (risk is less than 15%) for Coronary Heart Disease (CHD), fatal CHD, stroke and fatal stroke (the UKPDS Risk Engine provides risk estimates in individuals with type 2 diabetes not known to have heart disease (1), calculating the patient's risk involves considering risk factors such as age, sex, incidence of smoking and lipid levels)

Exclusion Criteria:

* Patients who do not meet the above criteria or are not willing to participate will not be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are type 2 diabetes patients who attend St.Paul's Diabetes Teaching and Training Centre (DTTC) and Dr. Hugh Tildesley's private office in Vancouver, BC Canada.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Tildesley, MD, Principal Investigator — St. Paul's Hospital, University of British Columbia
Locations (1):
- Endocrine Research Society, Vancouver, British Columbia, Canada